CLINICAL TRIAL: NCT01510470
Title: Clinical and Radiological Outcomes Study on Astra Tech Osseospeed Tx Profile Implant
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hong Kong Brånemark Osseointegration Center (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Dr. Philip Lee KM, Director, Hong Kong Brånemark Osseointegration Center, Hong Kong Brånemark Osseointegration Center
Other Study IDs: D2011028
Record Dates: First submitted 2012-01-11; First posted 2012-01-16 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Malocclusion; Displaced or Missing Teeth
Keywords: AstraTech Osseospeed Profile Implant; Marginal bone level; soft tissue; soft tissue responds
MeSH Terms: conditions — Malocclusion; Anodontia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Astra Tech Osseospeed Profile Implant design when placed in the healed extraction site maintains the marginal bone level

ELIGIBILITY:
Inclusion Criteria:

* Patients with single missing maxillary or mandibular premolar or molar
* The edentulous sites should be healed sites
* The opposing tooth will be a natural dentition

Exclusion Criteria:

* general contraindications to dental implant surgery
* Patient with irradiation in the head and neck region
* Immuno-suppressed or immuno-compromised patients
* Patients who took or are taking amino-bisphosphonates
* Patients with poor oral hygiene and motivation
* Patients with untreated periodontitis
* Uncontrolled diabetes
* Pregnancy or lactation
* Addiction to alcohol or other drugs
* patients with psychiatric problems
* Lack of occluding dentition/prosthesis
* Restricted mouth opening (less than 3.5cm inter-arch anteriorly)
* Patients with an acute or chronic infection/inflammation in the area intended for implant placement
* Patients unable to commit 5 years follow up
* Patients referred for implant placement only

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with single missing maxillary or mandibular premolar or molar
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Brånemark Osseointegration Centre, Hong Kong SAR, China